CLINICAL TRIAL: NCT06021873
Title: Evaluation of the Non-inferiority of the Robotic Approach Over the Laparoscopic Approach in Patients Who Are Candidates for Single Anastomosis Duodeno-ileal Bypass With Sleeve Gastrectomy (SADI-S)
Acronym: LvRSADIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5538
Record Dates: First submitted 2023-07-10; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-05

CONDITIONS: Obesity, Morbid
Keywords: minimally-invasive surgery; robotic surgery; single anastomosis duodeno-ileal bypass with sleeve gastrectomy (sadi-s)
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Monocentric, interventional, prospective, randomized 1:1, with comparison of two surgical approaches
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic SADI-S (Active Comparator): Patients with indication to laparoscopic Single-anastomosis duodeno-ileal bypass with sleeve gastrectomy
  Interventions: Procedure: SADI-S
- Robotic SADI-S (Active Comparator): Patients with indication to robotic Single-anastomosis duodeno-ileal bypass with sleeve gastrectomy
  Interventions: Procedure: SADI-S

INTERVENTIONS:
Procedure: SADI-S — Single-anastomosis duodeno-ileal bypass with sleeve gastrectomy

SUMMARY:
Treating patients with super-obesity has always been challenging for bariatric surgeons due to the higher risk of postoperative complications and the limited success of commonly used bariatric procedures (restrictive and hypo-absorptive). In this context, these patients are often considered for more complex procedures, such as hypo-absorptive interventions. Over the past 15 years, a new hypo-absorptive procedure called single-anastomosis duodenal switch with biliopancreatic diversion (SADI-S) has been introduced and recognized as a bariatric procedure by leading national and international scientific societies. It has shown promising short- and medium-term results regarding weight loss and metabolic improvements.

The SADI-S procedure is a technically complex multi-quadrant surgery. This study aims to evaluate the equivalence in terms of morbidity between laparoscopic and robotic approaches for patients undergoing this procedure.

DETAILED DESCRIPTION:
Patients with super-obesity (BMI≥50 kg/m2) present a significant challenge for bariatric surgeons due to the complexity of their cases. Hypo-absorptive procedures are often necessary to achieve the best results in weight loss and metabolic improvements. However, these procedures are known to be among the most difficult to perform, especially in super-obese patients. In recent years, there has been considerable interest in applying robotic technology to bariatric surgery, specifically for hypo-absorptive procedures.

The single-anastomosis duodenal switch with biliopancreatic diversion (SADI-S) has gained significant attention among the various hypo-absorptive procedures. This procedure is technically less complex than others, thanks to its reconstruction with a single anastomosis between the duodenum and the ileum. Despite its technical advantages, it maintains the original procedure's desired bariatric and metabolic outcomes. SADI-S is now recognized as an established bariatric procedure by major national and international scientific societies.

However, there is ongoing debate regarding the equivalency of laparoscopic and robotic approaches regarding complications, morbidity, and mortality. Thus, this study aims to evaluate the safety and effectiveness of both minimally invasive approaches (laparoscopic and robotic) in patients undergoing SADI-S.

The study will have a monocentric design involving a prospective, interventional, and randomized comparison between the two surgical strategies. The target population includes patients eligible for SADI-S using a minimally invasive technique, with inclusion criteria being age 18 years or older and informed consent. Patients eligible for different bariatric procedures be excluded.

The study will span a duration of 5 years, and the aim is to enroll an average of 105 patients per year to achieve the final sample size. Primary endpoints include comparing the risk of postoperative complications within 30 days of surgery between the laparoscopic and robotic approaches. Secondary endpoints encompass evaluating intraoperative complications, conversion rates, mortality, operative times, and post-operative hospital stay and conducting a cost analysis of both approaches.

However, there is ongoing debate regarding the equivalency of laparoscopic and robotic approaches in terms of complications, morbidity, and mortality. Thus, the objective of this study is to evaluate the safety and effectiveness of both minimally invasive approaches (laparoscopic and robotic) in patients undergoing SADI-S.

The study will have a monocentric design, involving a prospective, interventional, and randomized comparison between the two surgical strategies. The target population includes patients eligible for SADI-S using a minimally invasive technique, with inclusion criteria being age 18 years or older and informed consent. Patients eligible for different bariatric procedures be excluded.

The study will span a duration of 5 years, and the aim is to enroll an average of 105 patients per year to achieve the final sample size. Primary endpoints include comparing the risk of post-operative complications within 30 days of surgery between the laparoscopic and robotic approaches. Secondary endpoints encompass evaluating intraoperative complications, conversion rates, mortality, operative times, post-operative hospital stay, and conducting a cost analysis of both approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients eligible for Single-anastomosis duodeno-ileal bypass with sleeve gastrectomy using a minimally invasive technique
* Informed consent

Exclusion Criteria:

* Patients eligible for different bariatric procedures than SADI-S

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of post-operative complications | 30 days
  Comparison between the laparoscopic and robotic approach to Single-anastomosis duodeno-ileal bypass with sleeve gastrectomy in order to evaluate the post-operative complications rate within 30 days from the surgical procedure. Complications will be expressed in absolute numbers and divided into major complications (grade III-IV) and minor complications (grade I-II) according to the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Evaluation of morbidity, mortality and cost-analysis | 30 days
  Comparison between the laparoscopic and robotic approach to Single-anastomosis duodeno-ileal bypass with sleeve gastrectomy. Our evaluation focuses on: the rate and percentage of intra-operative complications, the conversion rate and percentage, operative time (expressed as 'skin-to-skin' time in minutes), the length of hospital stay (in days), and cost analysis. In Italy, bariatric surgery has a flat reimbursement rate of 5681.3€ regardless of the surgical method (laparoscopic or robotic) or postoperative complications. We will conduct a cost analysis combining bottom-up micro-costing and top-down gross costing. Specifically, operating room costs, which encompass anesthesia, surgery, and scrub nurse professionals, as well as utilities, will be calculated with top-down gross costing. Hospital stay costs will combine micro-costing for drugs and tests with top-down costing for surgical/nurse professionals and accommodation.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Raffaelli, Prof, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided